CLINICAL TRIAL: NCT04343144
Title: Cohort Multiple Randomized Controlled Trials Open-label of Immune Modulatory Drugs and Other Treatments in COVID-19 Patients CORIMUNO-19-Nivolumab Trial
Brief Title: Trial Evaluating Efficacy and Safety of Nivolumab (Optivo®) in Patients With COVID-19 Infection, Nested in the Corimmuno-19 Cohort.
Acronym: CORIMUNO-NIVO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200389-5
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: COVID19- Infection With SARS-CoV-2 Virus
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: 2 parallels arms randomized open-label multi center clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nivolumab (Experimental)
  Interventions: Drug: Nivolumab Injection
- Standard of Card (No Intervention)

INTERVENTIONS:
Drug: Nivolumab Injection — Treatment consists of an infusion of OPDIVO® 3mg/kg on day 1 (D1).
  Arms: Nivolumab

SUMMARY:
It appears interesting to use nivolumab in severe patients infected with SARS-CoV-2 requiring hospitalization in conventional unit or in ICU.

This protocol CORIMUNO19-NIVO therefore, will evaluate the efficacy and safety of OPTIVO® (nivolumab) COVID-19 patients hospitalized in conventional unit.

The purpose of this study is to show the efficacy of nivolumab in patients with COVID-19 in combination with standard treatments.

A phase 2 randomized open trial will evaluate the efficacy and safety of optivo® (nivolumab) alone versus standard of care (SoC) in patients hospitalized in conventional units.

Patients will be randomly allocated 1:1 to either nivolumab or SoC.

ELIGIBILITY:
Inclusion Criteria:

* Adults (men and women) age over 18 years old
* At least one nasal swab positive for COVID-19 detected by PCR, maximum 7 days prior to treatment
* Viral pneumonia confirmed by TDM scan
* Patients meeting all of the following 3 criteria:

  * Requiring more than 3L/min of oxygen
  * WHO progression scale = 5
  * No NIV or High flow

Exclusion Criteria:

* Patients with active cancer and immunocopromised patients
* Known hypersensitivity to nivolumab or to any of their excipients.
* Pregnancy
* Patient with an autoimmune or inflammatory disease (including but not limited to: Crohn's Disease, rheumatoid arthritis, scleroderma, systemic lupus erythematosus, Grave's disease). Patients with thyroiditis or vitiligo only could be included.
* Patient with a history of thymoma
* Patient with a history of solid organ transplantation or a bone marrow transplantation
* Patients treated with immune checkpoint inhibitors 3 months prior to the study
* Patients who had a history of grade 3 or 4 immune-related adverse events with a previous treatment with immune-checkpoint inhibtors
* Patients requiring ICU based on Criteria of severity of COVID pneumopathy
* Respiratory failure requiring mechanical ventilation or extracorporeal membrane oxygenation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Time to clinical improvement | day 14
  the time required for clinical improvement, defined as the time elapsed between randomization and a two-point improvement on an ordinal scale with seven categories (WHO scale), or the discharge alive from hospital, whatever occurred first

SECONDARY OUTCOMES:
Overall survival | day 28
Overall survival | day 90
Cumulative incidence of ICU admission | day 28
Length of hospital stay | day 90
Positive nasal PCR | day 7
Incidence of adverse events | day 28
Incidence of grade 3-4 adverse events | day 28
  according to CTC AE-4.03
World Health Organisation (WHO) progression scale | day 4, 7 and 14
  range, from 0 (healthy) to 10 (death)

CONTACTS AND LOCATIONS:
Locations (1):
- Pneumologie hôpital Tenon, Paris, France